CLINICAL TRIAL: NCT03261570
Title: Cardiovagal Baroreflex Deficits Impair Neurovascular Coupling and Cognition in Postural Tachycardia Syndrome
Brief Title: Cardiovagal Baroreflex Deficits Impair Neurovascular Coupling and Cognition in POTS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Julian Stewart, Professor of Pediatrics, New York Medical College
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1R01HL134674-01A1 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-08

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS); POTS; Orthostatic Intolerance
Keywords: Postural Orthostatic Tachycardia Syndrome (POTS); POTS; Orthostatic Intolerance; Digoxin; Pyridostigmine; Mestinon
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Pyridostigmine Bromide; Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pyridostigmine and Placebo (Active Comparator): Pyridostigmine 60mg by mouth one day and Placebo (Lactulose 50mg) by mouth on a different day
  Interventions: Drug: Pyridostigmine; Drug: Placebo
- Digoxin and Placebo (Active Comparator): Digoxin 0.5mg (500mcg) by mouth one day and Placebo (Lactulose 50mg) by mouth on a different day
  Interventions: Drug: Digoxin; Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — 60mg by mouth
  Other Names: Mestinon
  Arms: Pyridostigmine and Placebo
Drug: Digoxin — 0.5 (500mcg) by mouth
  Arms: Digoxin and Placebo
Drug: Placebo — Lactulose 50mg by mouth

SUMMARY:
Postural tachycardia syndrome (POTS), is the chronic form of orthostatic intolerance associated with excessive upright tachycardia, and occurs predominantly in young females (>85%). Among its most troubling symptoms are lightheadedness, fatigue, and decreased memory often called "brain fog" by patients. Task-related neurovascular coupling (NVC) links neural activity to an increase in CBF known as "functional hyperemia". Although memory task performance and NVC deteriorated with angle of tilt in POTS but not healthy controls, cerebral blood flow (CBF) remained similar to control. Instead, the investigators observed extensive narrow band low frequency (0.07-0.13 Hz) oscillations in BP (OBP) that entrained and amplified oscillations in CBF (OCBF). OBP and OCBF increased with tilt angle and caused impaired working memory and reduced functional hyperemia. The cardiovagal baroreflex couples BP to HR to buffer BP changes. The investigators hypothesize that the cardiovagal baroreflex becomes progressively impaired with orthostasis in POTS, but not in healthy volunteers, and accounts for OBP, OCBF, and loss of NVC; further, improving the baroreflex reduces OBP, OCBF and Brain Fog in POTS.

DETAILED DESCRIPTION:
Orthostatic intolerance is defined by debilitating upright symptoms that are relieved by sitting or lying. Symptoms include upright lightheadedness, fatigue, confusion, and decreased memory called 'Brain Fog' by patients. The most common chronic form is Postural Tachycardia Syndrome (POTS), characterized by excessive upright tachycardia without hypotension. Of note, >85% of POTS patients are female. The proposal that Brain Fog was caused by reduced cerebral blood flow (CBF) has been disproven, because graded incremental upright tilt failed to demonstrate difference in mean CBF compared to healthy volunteers. Nevertheless, memory task performance deteriorates with angle of tilt as does task-related neurovascular coupling (NVC), which links neural activity to an increase in CBF known as "functional hyperemia". The investigators have previously observed that large low frequency (0.07-0.13 Hz) oscillations in BP (OBP), which entrained and amplified oscillations in CBF (OCBF), increased with tilt angle and were associated with impaired working memory and reduced functional hyperemia.

The sympathetic baroreflex remains intact and HR is excessively increased in the absence of parasympathetic counterregulation. The cardiovagal baroreflex couples BP to HR to buffer BP changes. Large low frequency BP oscillations, representing a resonance within the sympathetic baroreflex loop, occur if there is central hypovolemia, an intact sympathetic baroreflex, and reduced parasympathetic buffering of BP by HR; conditions found in upright POTS. This leads to the following hypothetical paradigm:

↓Cardiovagal Baroreflex → ↑OBP → ↑↑OCBF → ↓NVC → ↓working memory. Therefore, in this application, the investigators hypothesize that the cardiovagal baroreflex is impaired in POTS while supine, becomes further impaired with orthostasis, and accounts for OBP, OCBF, and loss of NVC. Further, the investigators propose that improving the cardiovagal baroreflex improves hemodynamics and Brain Fog in POTS patients.

ELIGIBILITY:
Inclusion Criteria for POTS patients:

POTS patients referred for day to day orthostatic intolerance with greater than 3 symptoms for greater than 3 months and will have the diagnosis of symptomatic postural tachycardia made during a screening tilt table test :

* dizziness
* nausea and vomiting
* palpitations
* fatigue
* headache
* exercise intolerance
* blurred vision
* abnormal sweating heat.

Healthy control subjects:

* normal physical examination, and normal electrocardiographic and echocardiographic evaluations.
* Only those free from heart disease, and from systemic illness will be eligible to participate.
* This excludes patients with illnesses and disease states known to be associated with endothelial cell dysfunction such as diabetes, renal disease, congestive heart failure, systemic hypertension, acute and chronic inflammatory diseases, neoplasm, immune mediated disease, trauma, morbid obesity and peripheral vascular disease.

At the time of testing all patients and control subjects must refrain from vasoactive drugs for two weeks.

Exclusion Criteria for both POTS and healthy controls:

* An active medical condition that may explain the diagnosis
* A previous medical condition with undocumented resolution that may explain the diagnosis
* any systemic or overt structural, arrhythmic or myopathic cardiovascular disease
* any illnesses known to produce autonomic dysfunction such as diabetes, heart disease, renal disease, systemic hypertension, acute and chronic inflammatory diseases, neoplastic disease, immune mediated disease, major trauma and burns, morbid obesity and peripheral vascular disease will also be excluded.
* Cigarette smokers will be excluded.
* Past or present major psychiatric disorder
* Substance abuse within 2 years before onset of symptoms.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Cardiovagal Baroreflex during orthostatic stress | 1 year
  Cardiovagal Baroreflex during orthostatic stress in unmedicated POTS patients compared to unmedicated control subjects during each angle of incremental tilt. The unmedicated baroreflex measurement will be repeated in POTS patients to similar measurements after treatment with placebo, pyridostigmine or digoxin. Baroreflex measurements will be obtained using the standard "modified Oxford" technique.
Cognitive ability during orthostatic stress | 1 year
  . Cognitive ability during orthostatic stress in unmedicated POTS patients compared to unmedicated control subjects during each angle of incremental tilt. Cognitive ability will be repeated in POTS patients to similar measurements after treatment with placebo, pyridostigmine or digoxin. Cognitive ability will be assessed with a standard 2-Back test in which patients identify identical alphabetic characters appearing 2 characters before the current displayed character in a sequence of 29 characters.

SECONDARY OUTCOMES:
Cardiac output measure by inert gas breathing technique | 1 year
  Cardiac output measure by inert gas breathing technique. Cardiac output is the amount of blood pumped by the heart in one minute. The technique uses the Innocor system in which the relative levels of two inert gases - one blood soluble and one insoluble component - are measured over a few respirations (about 5 breaths or 15 seconds). The rate of disappearance of the soluble gas from the alveolar space is proportional to the flow of blood perfusing the lungs and equals the cardiac output.
Arterial blood pressure, and mean arterial pressure defined by the time average blood pressure over the cardiac cycle | 1 year
  Arterial blood pressure in mmHg over each cardiac cycle will be collected using finger photoplethysmography. The arterial pressure is reported as an aggregate of 3 extracted quantities: the systolic blood pressure which is the maximum blood pressure over a cardiac cycle; the diastolic blood pressure which is the minimum blood pressure over a cardiac cycle; and the mean blood pressure which is the average blood pressure over a cardiac cycle.
Heart rate | 1 year
systemic vascular resistance defined by the ratio of mean arterial pressure to cardiac output | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julian M. Stewart, M.D., Ph.D., Principal Investigator — New York Medical College
Locations (1):
- New York Medical College/Bradhurst building, Hawthorne, New York, United States